CLINICAL TRIAL: NCT01138748
Title: Prediction of the Effectiveness of Hypofractionated Radiation Therapy in Early Stage Lung Cancer by Bio-imaging and Biomarkers
Acronym: PEARL-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Nationaal Kankerplan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/205; LONG 10-01 (Other: University Hospital Ghent)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Inoperable Early Stage Non-small Cell Lung Cancer
Keywords: inoperable early stage non-small cell lung cancer; radiation therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation therapy (Experimental)
  Interventions: Radiation: hypofractionated radiation therapy

INTERVENTIONS:
Radiation: hypofractionated radiation therapy — hypofractionated radiation therapy

SUMMARY:
Surgical resection with mediastinal lymph node sampling is currently the therapy of choice for early stage (I-II) non-small cell lung cancer (NSCLC). Selected patients unwilling or unable to tolerate surgery are referred for so-called 'curative' high dose radiotherapy. This has shown to result in a long term local disease control rate and a high cancer specific survival.

The current trial addresses the issue if progression free survival (PFS) in patients treated with radiotherapy can be predicted by a multi-variate model derived from a composite of bio-imaging and biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Proof of cT1a/b - 2a/b N0M0 NSCLC
* Informed Consent signed
* Resectable tumour
* > 18 years old
* men and women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
development and validation of a multi-variate predictive model | from 2 to 5 years
  To develop and validate a multi-variate predictive model based on bio-imaging and biomarkers for progression)free survival from 2 to 5 years.

SECONDARY OUTCOMES:
the clinical response and complication rate | from 2 to 5 years
local, regional or distant failure | from 2 to 5 years
progression free survival | from 2 to 5 years
disease specific overall survival | from 2 to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Meerbeeck, MD,PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of University Hospital Ghent — http://www.uzgent.be